CLINICAL TRIAL: NCT01783457
Title: e-Learning & Development of an Evidence-based Psychoeducational Programme for First Episode Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Ana María González-Pinto, Ph.D. in Medicine, Psychiatrist, Lecturer at University of the Basque Country, Chief of Psychiatry Department at Araba University Hospital, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PsychEd-FEP
Record Dates: First submitted 2013-01-23; First posted 2013-02-05 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Psychosis
Keywords: First psychotic episode; Individual psychoeducation; Telemedicine; BDNF; Oxidative stress
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual psychoeducation (Experimental): Usual treatment + individual psychoeducational intervention (14 sessions). The psychoeducational programme consists of 14 sessions of 60 minutes every other week for six months, focused on improving patient awareness of their condition, adherence to treatment, identification of prodromes, early intervention in potential relapses, anxiety management techniques, social skills, healthy lifestyle habits and problem solving.
  Interventions: Other: Individual psychoeducation
- Control (Active Comparator): Usual treatment
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — Usual treatment: pharmacological treatment + regular sessions with their psychiatrist.
  Other Names: Usual treatment
  Arms: Control
Other: Individual psychoeducation — Usual treatment + individual psychoeducational programme, consisting of 14 sessions of 60 minutes every other week for six months, focused on improving patient awareness of their condition, adherence to treatment, identification of prodromes, early intervention in potential relapses, anxiety management techniques, social skills, healthy lifestyle habits and problem solving.
  Programme of sessions available upon request.
  Arms: Individual psychoeducation

SUMMARY:
Treatment delay in psychosis usually lead to slower recovery, an increase in associated comorbidity and greater deterioration in social and family life of patients. Previous studies indicate that an early intervention with guidelines for increasing adherence to treatment, disease awareness and condition management leads to better progression of the disorder and is therefore related to a better prognosis.

Several studies have found that the rate of relapse is higher in patients with pharmacological treatment alone compared to those also receiving psychoeducation, who tend to improve their adherence to treatment and reduce toxic drugs dosage.

Hypotheses:

* Individual psychoeducation will be effective as complementary therapy to pharmacological treatment in patients with a first psychotic episode, improving disease evolution.
* BDNF levels will increase more in the patients receiving individual therapy compared to those without it.
* Psychoeducation can be performed similarly in all participating centers if the therapists receive the same training and use the same psychoeducation material.
* The use of telemedicine for the follow-up of the patients will help improve the welfare work and therefore the disease evolution.

DETAILED DESCRIPTION:
Treatment delay in psychosis usually lead to slower recovery, an increase in associated comorbidity and greater deterioration in social and family life of patients. Previous studies indicate that an early intervention with guidelines for increasing adherence to treatment, disease awareness and condition management leads to better progression of the disorder and is therefore related to a better prognosis.

Several studies have found that the rate of relapse is higher in patients with pharmacological treatment alone compared to those also receiving psychoeducation, who tend to improve their adherence to treatment and reduce toxic drugs dosage.

Hypotheses:

* Individual psychoeducation will be effective as complementary therapy to pharmacological treatment in patients with a first psychotic episode, improving the disease evolution.
* BDNF levels will increase more in the patients receiving individual therapy compared to those without it.
* Psychoeducation can be performed similarly in all participating centers if the therapists receive the same training and use the same psychoeducation material.
* The use of telemedicine for the follow-up of the patients will help improve the welfare work and therefore the disease evolution.

Primary Objective:

* To assess the effectiveness of individual psychoeducation together with telemedicine (telephone assistance) as an adjuvant therapy in the pharmacological treatment of patients with first episode psychosis, regarding functionality of patients and positive and negative symptoms.

Secondary Objectives:

* To analyse certain biological parameters (BDNF and oxidative stress) in both arms (intervention and control) at baseline and during re-assessment (at six months and after completion of treatment).
* To analyse the effectiveness of online training of psychotherapists who will provide psychoeducation to patients with first episode psychosis.

ELIGIBILITY:
Inclusion Criteria:

* patients who have suffered a first psychotic episode (diagnosis IV-TR) in the last five years,
* age between 18 and 45 years,
* patients who have given written informed consent to participate.

Exclusion Criteria:

* patients with a comorbid disorder that interferes with their ability to communicate,
* patients who received psychoeducation previous to inclusion in study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Prognosis of patients. | 6 months
  To assess the prognosis of patients by registering the number of relapses and the number of psychiatric hospital admissions.

SECONDARY OUTCOMES:
Score on clinical scales assessing functionality. | 6 months
  To assess the effectiveness of individual psychoeducation together with telemedicine (telephone assistance) as an adjuvant therapy in the pharmacological treatment of patients with first episode psychosis, using different scales for clinical assessment of FUNCTIONALITY (Positive and Negative Syndrome Scale (PANSS), SUMD, Morisky-Green Scale, STAI, Hamilton Rating scale for Depression, LSAS, WHOQOL-BREF, EuroQoL) and PROGNOSIS (Strauss Carpenter Scale, GAF, Functional Assessment Staging Test-FAST).
Score of participating psychotherapists on a specific test after online training. | 6 months
  To analyse the effectiveness of online training of psychotherapist who will provide psychoeducation to patients, all therapists carried out a specific tests after each one of the sessions to confirm if they had delivered the session as specified in the protocol.
Biological Parameters: blood levels of BDNF. | 6 months
  To analyse BDNF biological parameter at baseline and during re-assessment at six months (after completion of treatment): BDNF levels in plasma will be measured by ELISA techniques with a kit based on the Sandwich technique used according to the manufacturer´s instructions (CYT306 from Chemicon). The standard curves will be characterised using plasma duplicates and the absorption determined with a microplate reader (BIO-TEK, Sinergy HT) using a wavelength of 450 nm.
Biological Parameters: levels oxidative stress indicators in blood. | 6 months
  To analyse OXIDATIVE STRESS indicators at baseline and during re-assessment at six months (after completion of treatment): Levels of the following OXIDATIVE STRESS INDICATORS will be measured in red blood cell haemolysates: lipid peroxidation (TBARS), nitrites and superoxide dismutase enzyme, total antioxidant ability, glutathione peroxidase and catalase.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Vega, Psychologist, Study Chair — Santiago Hospital - Basque Health Service
Locations (6):
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Hospitalet Llobregat, Barcelona
  - Fundación Clínico Valencia INCLIVA, Valencia, Valencia
  - Universidad de Valencia, Valencia, Valencia
  - Universidad del País Vasco, Bilbao, Vizcaya
  - Araba University Hospital-Santiago, Vitoria-Gasteiz, Álava

REFERENCES:
- [Derived] Barbeito S, Vega P, Ruiz de Azua S, Balanza-Martinez V, Colom F, Lorente E, Luengo A, Cerrillo E, Crespo JM, Gonzalez Pinto A. Integrated treatment of first episode psychosis with online training (e-learning): study protocol for a randomised controlled trial. Trials. 2014 Oct 27;15:416. doi: 10.1186/1745-6215-15-416. PMID 25348346